CLINICAL TRIAL: NCT04317001
Title: Developing Improved Treatment for Cognitive Impairment in Depression
Brief Title: Treatment for Cognitive Impairment in Depression
Acronym: T-CID
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Researcher leading the study moved institutions study not feasible
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Leanne Williams, Professor, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 46217
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Major Depressive Disorder
Keywords: cognition
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active treatment with modafinil (Active Comparator): active intervention
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): placebo intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Treatment will be with 100mg of modafinil for the two week primary phase of the study
  Other Names: Provigil
  Arms: Active treatment with modafinil
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The proposed study seeks to investigate the effects of modafinil on cognitive function in depression, which holds promise for better treating cognitive impairment in depression, as well as better understand cognitive dysfunction in MDD from a neural rather than diagnostic point of view to better classify and treat these disabling symptoms.

DETAILED DESCRIPTION:
Vortioxetine is the only FDA approved medication for treating cognitive impairment in depression. This medication, however, takes a minimum of 6-8 weeks to take effect and is only effective in a subset of patients. Modafinil, has shown some benefit in off-label treatment of cognitive dysfunction in psychiatric disorders. The effects of modafinil on cognitive function in both healthy controls and treatment resistant and partially remitted individuals with MDD have shown promising results. To date, however, studies have focused on modafinil's potential as an augmenting agent for treatment resistant depressive symptoms, but have not examined its effects on cognitive function in depression as a primary outcome measure. Modafinil's ability to treat cognitive symptoms in non-treatment refractory or partially remitted individuals specifically struggling with cognitive impairment resulting from MDD have not been assessed. Further, we lack a mechanistic understanding of modafinil's effects on brain circuitry.

The proposed research seeks to examine the effects of modafinil on different domains of cognitive function such as attention, working memory and processing speed, as well as its underlying effects on brain circuitry in individuals who demonstrate cognitive impairment and meet criteria for first episode of major depressive disorder. Specifically, this study would examine the effect of administering low dose modafinil, a drug that has been used off-label to treat cognitive dysfunction in psychiatric disorders, on cognitive function in major depressive disorder in a two-session double-blind, randomized, placebo-controlled design.

The primary aim of the study is to examine the effect of modafinil on domains of cognitive processing and function in depression as well as the neural mechanisms underlying its effects using functional magnetic resonance imaging (fMRI). A secondary aim of this study is to compare the efficacy of modafinil in treating cognitive dysfunction to that of vortioxetine in an optional phase 2 open-label follow up. In an optional second phase of the study, participants randomized to the placebo group, will have the option of enrolling in an open label trial of either modafinil or vortioxetine, the only currently FDA approved medication to treat cognitive impairment in depression. Study findings may provide the foundations for future work focused on treating cognitive impairment in depression.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age (inclusive)
* Fluent and literate in English, and show non-impaired intellectual abilities to ensure adequate comprehension of the task instructions
* Meet diagnostic criteria for major depressive disorder
* Experiencing cognitive impairment attributed to depression that perform less than 0.5 standard deviations below the norm on a minimum of two cognitive domains on baseline cognitive testing
* Medication naïve to Modafinil. (Subjects can previously have been treated on antidepressants. If their usual treating physician is supportive, participants who are currently on an antidepressant can be tapered off the antidepressant to participate.)
* Written, informed consent
* MRI scanning eligibility, including no evidence of any form of metal embedded in the body (e.g., metal wires, nuts, bolts, screws, plates, sutures), as these produce artifacts when brain imaging. All potential subjects will need to successfully complete the screening forms at the Stanford Center for Cognitive and Neurobiological Imaging (CNI).

Exclusion Criteria:

* Current Axis 1 psychiatric disorder other than major depressive disorder
* Concurrent participation in other intervention or treatment studies
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with ability to complete the assessments, or are unable and/or unlikely to follow the study protocols
* Impaired decision-making capacity
* Medical/neurological illness that result in cognitive impairment
* Current or prior use of psychotropic medications
* Body Mass Index outside healthy range (18-30).
* Magnetic resonance contraindication
* History of alcohol or substance (e.g., sedative-hypnotics, cannabis, stimulants, opioids, cocaine, hallucinogens) abuse or dependence
* Lifetime history of medical illness that may compromise cognitive functioning (including neurological disorders such as seizures or stroke, Parkinson's disease, dementia)
* History of head injury with loss of consciousness
* History of mental retardation
* Active suicidal ideation or history of suicide attempt in past year
* Treatment-resistant hypertension or any known cardiovascular disease
* Women who are pregnant or breastfeeding
* Kidney or liver function impairment
* Taking any medication contraindicated with modafinil including hormonal contraceptives, anticonvulsants (e.g. diazepam, phenytoin), propranolol, warfarin, drugs that are metabolized by CYPC19 or CYP3A enzymes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress Scale (DASS) | Day 1, Day 14 and Day 28
  A 42-item self report scale that can be considered in the context of depression using the DASS depression scale.

IPD SHARING:
Plan to Share IPD: No